CLINICAL TRIAL: NCT02423785
Title: Exploratory Study Investigating Ocular Blood Flow in Colorectal Cancer Patients Before and After Treatment With Anti-angiogenic Therapy
Brief Title: Ocular Blood Flow in Colorectal Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thorsten Fuereder, Dr.med., Medical University of Vienna
Other Study IDs: OBF-13
Record Dates: First submitted 2014-07-31; First posted 2015-04-22 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In colorectal cancer therapy anti-angiogenic strategies have become a cornerstone of treatment regimens in the metastatic setting. Addition of bevacizumab to conventional chemotherapeutic combination regimens has improved the median overall survival of advanced colorectal cancer patients by approximately 5 months. Selecting patients, who will benefit from anti-angiogenic approaches, would be highly desirable in order to optimize treatment strategies. Changes in ocular blood flow may be an attractive biomarker for predicting treatment response. In light of the given alternative first line treatment options such a predictive biomarker would be of clinical benefit. In the proposed study the investigators will assess potential changes in the ocular blood flow of mCRC patients after treatment with standard of care anti-angiogenic/cytotoxic therapy as an early predictive marker of treatment response as assessed by standard CT-scan

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (age 18 and over) suffering from mCRC.
* Normal findings in ophthalmic examination (except the investigator finds an abnormality irrelevant for the purpose of the study.)
* Patients, which are scheduled for standard of care treatment with chemotherapy plus bevacizumab

Exclusion Criteria:

* Refusal to give informed consent
* Severe hypertension (RR ≥180/110)
* Epilepsy
* Pregnancy and breastfeeding women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who are treated at the Medical University of Vienna
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-05; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Correlation between ocular blood flow (retinal blood flow) and treatment response | Within 2-3 months at restaging
  mean RBCs velocity in Hz and blood flow in arbitrary units will be reported and correlated with response rates (CR,PR,SD or PD)
Correlation between retinal vessel diameter and treatment response | Within 2-3 months at restaging
  Retinal vessel diameter will be reported and correlated with response rates (CR,PR,SD or PD)
Changes in retinal surface before and after therapy as measured by optical coherence tomography | Within 2-3 months at restaging

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria